CLINICAL TRIAL: NCT04187365
Title: Optimizing the Management of Postpartum Urinary Retention: Postpartum Urinary Retention (PUR) Study
Brief Title: Optimizing the Management of Postpartum Urinary Retention
Acronym: PUR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated prematurely due to challenges with recruitment and feasibility of continuing the study
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Sarah Collins, Assistant Professor, Department of Obstetrics & Gynecology, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00210382
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Urinary Retention
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Intervention Model Description: In Arm 2, women with severe postpartum urinary retention will be randomized to 3 or 7 days of foley catheter.
Masking Description: No masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP 1 (NonSevere PUR and women without PUR) (No Intervention): Women in GROUP 1 will be prospectively observed to characterize their clinical outcomes.
- GROUP 2 (Severe PUR) (Experimental): Women in GROUP 2 will be a randomized to either 3 or 7 days of indwelling catheterization.
  Interventions: Other: Duration of Indwelling Catheter

INTERVENTIONS:
Other: Duration of Indwelling Catheter — Foley catheter
  Arms: GROUP 2 (Severe PUR)

SUMMARY:
A study aimed at characterizing the comparing duration of catheterization for treatment of postpartum urinary retention (PUR) and characterizing short and long-term pelvic floor symptoms in women who have PUR.

DETAILED DESCRIPTION:
The purpose of the study is to compare clinical outcomes of women with bladder distension injuries due to postpartum urinary retention (PUR) who have varying duration of catheterization for initial treatment of postpartum urinary retention.

Hypotheses

1. Longer duration of therapeutic catheterization will be associated with resolution of postpartum voiding dysfunction in women who sustain severe bladder distension injuries due to postpartum urinary retention.

   Definition of resolution of postpartum voiding dysfunction:

   A. A post void residual volume of less than half of initial instilled volume on the first retrograde voiding trial, AND B. No need for re-treatment for urinary retention within 1 week
2. The incidence of postpartum urinary retention (PUR) will vary by route of delivery, with operative vaginal delivery having the highest incidence.
3. Risk factors for PUR will be related to intrapartum and delivery conditions

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18.
2. Vaginal or cesarean delivery at term (37 weeks gestational age or later) of live-born infants.
3. English or Spanish speaking and reading.

Exclusion Criteria:

1. Adults unable to consent.
2. Women under the age of 18.
3. Women who are currently pregnant (All women in the study will have already delivered).
4. Prisoners or detained individuals.
5. Women who chronically use a urinary catheter for another medical condition.
6. Women with a neurological disease with bladder manifestations (examples: Cerebrovascular accidents, Multiple sclerosis, Parkinson disease, cerebral palsy).
7. Women with preeclampsia requiring magnesium treatment for seizure prevention.
8. Women with prior PUR
9. Women on anticholinergic medications.
10. Women who are actively being treated for a UTI.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2022-02-27 (Actual); Study Completion 2022-02-27 (Actual)

PRIMARY OUTCOMES:
To evaluate whether 3 days of indwelling catheterization is inferior to 7 days in resolving postpartum urinary retention. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Collins, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No